CLINICAL TRIAL: NCT01365858
Title: Effectiveness of Virtual Reality-based Cognitive Training in Daily Living in Stroke Patients Using Virtual Action Planning Supermarket (VAP-S)
Brief Title: Virtual Action Planning in Stroke: a Control Rehabilitation Study
Acronym: VAPS REHAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: CHUBX 2009/25
Record Dates: First submitted 2011-05-30; First posted 2011-06-03 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Virtual reality-based cognitive training (Experimental)
  Interventions: Other: Rehabilitation
- Cognitive rehabilitation (without extra computer training) (Active Comparator)
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — The experimental group patients receive rehabilitation by training "Virtual Action Planning - Supermarket" on a computer 45 minutes 5 times a week during a 2-week period. The control group will receive similar duration cognitive rehabilitation (no extra computer training) during this period (problem solving and occupational therapy).

SUMMARY:
* Background : The general experience with the Virtual Reality application approach suggests that this treatment concept is promising in stroke rehabilitation
* Purpose : In shopping activity in a real supermarket and in simulated with the investigators virtual shopping simulation (VAP-S = virtual action planning supermarket), the investigators will compare people who had undergone a stroke who receive conventional rehabilitation or virtual training in VAP-S.

DETAILED DESCRIPTION:
The objective of this study is firstly to examine the effectiveness of using virtual reality-based training VAP-S on the ability to run errands in a real supermarket in individuals with stroke. Virtual environment provide useful way to explore planning and secondly to examine the effectiveness of using VR in the assessment of cognitive planning for patients. A virtual supermarket was designed in which participants carried out a task close to daily activities: a test of shopping list. Of the 70 subjects (7 centres), 35 randomly allocated to the control group, and the other 35 subjects randomly allocated to the experimental group. Subjects will be evaluated by a therapist who will not be involved in the training program and did not know about the subject's group assignment.

Statistical analysis : We will calculate descriptive statistics for the clinical characteristics of each group. We will use to compare the baseline demographic characteristics, the pretraining and posttraining variables between groups, independent-samples t-tests for means and Chi-square tests for frequencies. A significance level of 0.05 is set for all analyses.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* 1 to 18 months after stroke
* Without dementia or previous clinical stroke
* With executive impairment (Grefex battery)
* Barthel score equal or more than 40
* With cognitive disability leading to specific rehabilitation
* Given and informed consent

Exclusion Criteria:

* dementia or severe psychiatric disease
* epilepsy
* disorder of consciousness
* visual agnosia
* severe visual impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-05; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Ability to perform shopping test in real supermarket (all items collected and all actions needed done) | After rehabilitation (day 16)

SECONDARY OUTCOMES:
Time to perform all actions in real shop; performance in virtual shopping simulation (number of items, time, inappropriate actions); user and caregiver satisfaction. | Before (day 1) and after (day16) rehabilitation

CONTACTS AND LOCATIONS:
Overall Officials: Geneviève CHENE, Pr, Study Chair — University Hospital, Bordeaux; Pierre-Alain JOSEPH, Pr, Principal Investigator — University Hospital, Bordeaux
Locations (7):
- France (7):
  - CHU Bordeaux, Bordeaux
  - Ap-Hp Garches, Garches
  - Hospices Civils de Lyon, Lyon
  - Chu Nancy, Nancy
  - Centre Mutualiste Rééducation et de Réadaptation Fonctionnelle de Kerpape LORIENT, Ploemeur
  - Chu Rennes, Rennes
  - Chu Saint-Etienne, Saint-Etienne